CLINICAL TRIAL: NCT06067659
Title: Comparison Of The Treatment Effects Of Extracorporeal Shockwave Therapy And Kinesiological Banding In Patients With Calcaneal Spur
Brief Title: Comparison Of The Treatment Effects Of Different Methods In Patients With Calcaneal Spur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Lecturer, University of Beykent
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UBeykent-5
Record Dates: First submitted 2023-09-04; First posted 2023-10-05 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Heel Spur
Keywords: Extracorporeal Shock Wave Therapy; Heel Spur; Kinesio Taping
MeSH Terms: conditions — Heel Spur | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Factorial Assignment randomized controlled trial 3 groups
Who Masked: Participant
Masking Description: Inclusion criteria for the study were diagnosis of calcaneal spur by a physician, being in the age range of 30-70 years, patient complaining of pain in the heel region, appearance of calcaneal protrusion in the radiographic image, no other treatment or medication (NSAI, steroids, other drugs, etc.) analgesics) and the patient volunteered to participate in the study. Exclusion criteria were those who received injection therapy to the foot area (corticosteroids or corticosteroids/anesthetics), those with a history of rheumatic disease, coagulopathy, thrombophlebitis, neoplasia, systemic inflammatory disease, and outpatient surgery in the last 3 months. No other treatment or medication (NSAI, steroids, other analgesics) will be used during the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Extracorporeal shock wave therapy (Experimental): ESWT (EMS Swiss DolorClast® Classic) application will be applied to patients in groups 1 and 3 with a frequency of 15 Hz, a 2000 shock wave and an energy density of 2.5 bar. In practice, patients will be asked to lie in the prone position and keep the knee and hip joints in a neutral position. By placing a towel roll under the ankle, the heel will be stabilized to be applied. Using the ultrasound gel as an intermediate, the ESWT device will be applied to the medial part of the calcaneus.
  Interventions: Other: Extracorporeal shock wave therapy
- Group B: Kinesiology taping (Experimental): The material used in the taping will be 5 cm wide and 0.5 mm thick Kinesio® Tape. In practice, the patients were placed in the prone position and the ankle would be dorsiflexed at 10 degrees, and the band would be divided into 4 equal parts on the metatarsals of the 1/3 of the foot from the cruis, starting from the calcaneus. Then, taping will be performed from the medial to the lateral of the calcaneus, passing over the area where the pain is intense. Patients will be asked not to remove the applied tape for 3 days.
  Interventions: Other: Kinesiology taping
- Group C: Extracorporeal shock wave therapy+Kinesiology taping (Experimental): Patients in this group will be treated with both extracorporeal shock wave therapy and kinesiotape.
  Interventions: Other: Extracorporeal shock wave therapy; Other: Kinesiology taping; Other: Extracorporeal shock wave therapy+Kinesiology taping

INTERVENTIONS:
Other: Extracorporeal shock wave therapy — ESWT (EMS Swiss DolorClast® Classic) application will be applied to patients in groups 1 and 3 with a frequency of 15 Hz, a 2000 shock wave and an energy density of 2.5 bar. In practice, patients will be asked to lie in the prone position and keep the knee and hip joints in a neutral position. By placing a towel roll under the ankle, the heel will be stabilized to be applied. Using the ultrasound gel as an intermediate, the ESWT device will be applied to the medial part of the calcaneus.
  Other Names: GRUP A
  Arms: Group A: Extracorporeal shock wave therapy; Group C: Extracorporeal shock wave therapy+Kinesiology taping
Other: Kinesiology taping — The material used in the taping will be 5 cm wide and 0.5 mm thick Kinesio® Tape. In practice, the patients were placed in the prone position and the ankle would be dorsiflexed at 10 degrees, and the band would be divided into 4 equal parts on the metatarsals of the 1/3 of the foot from the cruis, starting from the calcaneus. Then, taping will be performed from the medial to the lateral of the calcaneus, passing over the area where the pain is intense. Patients will be asked not to remove the applied tape for 3 days.
  Arms: Group B: Kinesiology taping; Group C: Extracorporeal shock wave therapy+Kinesiology taping
Other: Extracorporeal shock wave therapy+Kinesiology taping — Patients in this group will be treated with both extracorporeal shock wave therapy and kinesiotape.
  Arms: Group C: Extracorporeal shock wave therapy+Kinesiology taping

SUMMARY:
Calcaneal spur (heel spur) is one of the most common disorders associated with foot pain. Patients may complain of pain at every step during the day, so it is important to find the most effective treatment method for patients. The aim of this study is to compare the therapeutic efficacy of extracorporeal shock wave therapy (ESWT) and kinesiology taping (KB) in patients with calcaneal spurs.

Thirty patients with calcaneal spurs will be included in the study. The gender, age, body weight, height, body mass index, and affected side of the patients will be recorded. Patients will be randomly divided into three treatment groups: ESWT to the first group, KB therapy to the second group, and combined ESWT+KB to the third group. Each group will be treated for five sessions, once a week for five weeks. ESWT 15Hz frequency will be applied as 2.5 Barr energy and 2000 Shock/session. It will be applied with the KB I and fan method and the tape will not be removed for three days after the application. In the pre- and post-treatment evaluations of the patients, heel sensitivity and sensory perception will be evaluated with the Foot structure Foot Posture Index (API). Visual Analog Scale (VAS), Quality of Life Short Form-36 (SF-36), Foot Function Index (AFI) and Windlass Test will be used.

DETAILED DESCRIPTION:
One of the most common pathologies that causes foot pain, negatively affects the individual's walking and reduces the quality of life is calcaneal spur (heel spur). Calcaneal spurs are fibro-cartilaginous protrusions varying in size that form around the calcaneal bone, the strongest, most important and rearmost bone in the foot.

Treatment aims to reduce pain, reduce inflation, and shrink and eliminate the spur. Conservative treatment includes exercises, massage, ultrasound, phonophoresis, laser, short wave diathermy, cryotherapy and extracorporeal shock wave therapy (ESWT) as physiotherapy applications.

ESWT are pressure waves delivered to the body to stimulate soft tissue growth through local hyperemia, neovascularization, reduction of calcification, inhibition of pain receptors and denervation to provide pain relief and healing of chronic processes. ESWT is also used effectively in the treatment of calcaneal spur.

The aim of this study is to observe the superiority, if any, of ESWT and KB in the treatment of each other or to show how effective the combined application of the two is in the treatment of calcaneal spur.

This study will be a single-blind, randomized controlled trial to compare the effectiveness of BP and ESWT in patients with calcaneal spurs. All procedures used will be carried out in accordance with the ethical rules of the Declaration of Helsinki and were approved by the Amasya University Clinical Research Ethics Committee (E-30640013-050.01.04-126508). The study will be carried out on patients who applied to the Physical Therapy and Rehabilitation Polyclinic of a hospital between 10.10.2023 and 10.12.2023 with the complaint of heel pain and diagnosed with calcaneal spur.

Inclusion criteria for the study were diagnosis of calcaneal spur by a physician, being in the age range of 30-70 years, patient complaining of pain in the heel region, appearance of calcaneal protrusion in the radiographic image, no other treatment or medication (NSAI). , steroids, other drugs, etc.) analgesics) and the patient volunteered to participate in the study. Exclusion criteria were those who received injection therapy to the foot area (corticosteroids or corticosteroids/anesthetics), those with a history of rheumatic disease, coagulopathy, thrombophlebitis, neoplasia, systemic inflammatory disease, and outpatient surgery in the last 3 months. No other treatment or medication (NSAI, steroids, other analgesics) will be used during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of calcaneal spur by the physician
* Be between 30-70 years old
* The patient complains of pain in the heel region
* Appearance of the calcaneal protrusion on the radiographic image
* Not taking any other treatment or medication (NSAI, steroids, other analgesics) until 4 weeks before the start of the study.
* The patient's willingness to participate in the study.

Exclusion Criteria:

* Those who received injection therapy to the foot area in the last 3 months (corticosteroids or corticosteroids/anesthetics),
* Those with rheumatic disease, coagulopathy, thrombophlebitis, neoplasia history, systemic inflammatory disease
* Those with a history of outpatient surgery

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Day 1 and 5 weeks later
  It is a subjective evaluation method that converts some values that cannot be measured numerically into numbers. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line (no pain at all, I have excruciating pain) and the patient will be asked to indicate where on this line their situation is appropriate by drawing a line or pointing or pointing.
Foot Function Index | Day 1 and 5 weeks later
  It is a self-filled form developed to measure the effects of foot pathologies on pain, disability and activity limitation. Foot function index; It consists of 23 items with 3 subgroups as pain, disability and activity limitation. A higher score indicates more pain, disability, and activity limitation.

SECONDARY OUTCOMES:
Sociodemographic information | Day 1 and 5 weeks later
  Participants' age will be recorded in years, height in centimeters, body weight in kilograms, gender in male and female, and affected side in left and right.
Quality of Life Short Form-36 | Day 1 and 5 weeks later
  It is a thirty-six-question questionnaire that asks questions about the quality of daily life and the general health of the person, including how he or she has been feeling lately. SF-36 consists of 36 items assessing nine subscales. Evaluation: Each of the 36 items is given a score between 0 and 100, depending on the answers. The higher the score, the better the quality of life It means at a high level.
Windlass Test | Day 1 and 5 weeks later
  The plantar fascia is stretched when a load is present on the sole of the foot. The medial longitudinal arch is stretched to create more than 20 degrees of extension in the tarsal bones, and with it, a tensile force occurs in the plantar fascia. It is aimed to further stretch the fascia by extending the toes while the sole of the foot is in contact and the plantar fascia is taut. On physical examination, there is tenderness with finger pressure around the medial calcaneal tubercle, which is the attachment point of the plantar fascia to the calcaneus. When the thumb is forced into dorsiflexion, the plantar fascia will be stretched, causing pain at the attachment point of the fascia to the calcaneus. This is known as the windlass test.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin şAHBAZ, Study Director — İstanbul Beykent Üniversitesi
Locations (1):
- Yasemin ŞAHBAZ, Beyli̇kdüzü, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No